CLINICAL TRIAL: NCT01838785
Title: Positron-Emission Tomography With Vesicular Monoamine Transporter Ligand ([18F]-DTBZ) In Healthy Elderly And Young Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 99-4149A
Record Dates: First submitted 2013-04-21; First posted 2013-04-24 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2016-01

CONDITIONS: Healthy
Keywords: 18F-DTBZ AV-133 imaging
MeSH Terms: interventions — florbenazine F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-DTBZ AV-133 (Experimental): 18F-DTBZ AV-133 imaging
  Interventions: Drug: 18F-DTBZ AV-133

INTERVENTIONS:
Drug: 18F-DTBZ AV-133

SUMMARY:
A total 25 healthy subjects will be included in this study. Subjects between 20 and 80 years of age may be eligible for this study. Candidates are screened with a medical history and physical examination, and blood test.

DETAILED DESCRIPTION:
The primary objective of this protocol is to assess the possible age-dependent decline in striatal 18F-DTBZ uptake of healthy subjects.

This study is expected to be completed in a period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 20 years to 80 years.
2. Subjects without significant neuropsychiatric disorder after evaluation by Neurologist.
3. Subjects who provide a written informed consent prior to study entry. If the subject is incapable of informed consent, the caregiver may consent on behalf of the subject (the subject must still confirm assent).

Exclusion Criteria:

1. Pregnancy and breast feeding.
2. Significant recent (within 6 months) history of neurological (including stroke and brain trauma) or psychiatric disorder.
3. Alcohol or substance abuse within last year.
4. Parkinson's disease or other brain degenerative disease (spinocerebellar ataxia, Wilson's disease, hydrocephalus, multiple infarction, history of severe head injury or intracranial operation.
5. Unable to stay still in the MRI or PET scanner for 30 minutes.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- 18F-DTBZ AV-133: 18F-DTBZ AV-133 imaging
  18F-DTBZ AV-133
Period: Overall Study
Arm/Group | 18F-DTBZ AV-133
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 18F-DTBZ AV-133
Number analyzed (Participants) | 25
Age, Customized [Number; unit: participants]
  20-29 years | 5
  30-39 years | 6
  40-49 years | 7
  50-59 years | 4
  >60 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Region of Enrollment [Number; unit: participants]
  Taiwan | 25

OUTCOME MEASURES:

1. Primary Outcome: Age-Dependent Change in Striatal 18F-DTBZ Uptake of Healthy Subjects.
Time Frame: two years
Measure: Mean (95% Confidence Interval); unit: SUVR
Arm/Group | 18F-DTBZ AV-133
Number analyzed (Participants) | 25
SUVR | 0.05 [0.05 to 1.00]

2. Secondary Outcome: The Test/Retest 18F-DTBZ PET Measurements of VMAT2 Binding in Healthy Subjects.
Time Frame: two years
Population: A subgroup of 5 subjects receive additional scan for a test/retest reliability study
Measure: Mean (80% Confidence Interval); unit: SUVR
Arm/Group | 18F-DTBZ AV-133
Number analyzed (Participants) | 5
SUVR | 2.35 [1.18 to 3.94]

ADVERSE EVENTS:
Time Frame: one month
Arm/Group | 18F-DTBZ AV-133
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No